CLINICAL TRIAL: NCT06148662
Title: The Effect of Oral Sprays on Salivary pH Changes After Coca-cola Consumption
Brief Title: The Effect of Oral Sprays on Salivary pH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 18081215
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-11

CONDITIONS: Oral Health
Keywords: Coca-cola; salivary buffer capacity; salivary pH; oral foams
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No intervention (negative control) (Experimental): Negative control
  Interventions: Other: No intervention (negative control)
- Water (positive control) (Experimental): Tap water
  Interventions: Other: Water (positive control)
- Dental foam "Biorepair PERIBIOMA" (Experimental): Ingredients:
  Aqua, Sorbitol, Xylitol, Zinc Hydroxyapatite, Aroma, Pistacia Lentiscus (Mastic) Gum Oil, Lactobacillus, Bifidobacterium, Sodium Hyaluronate, Ascorbic Acid, Hamamelis Virginiana Leaf Extract, Spirulina Platensis Extract, Calendula Officinalis Flower Extract, Tocopheryl Acetate, Retinyl Palmitate, Eucalyptus Globulus Leaf Oil, PEG-40 Hydrogenated Castor Oil, Phenoxyethanol, Sodium Benzoate, Cocamidopropyl Betaine, Glycerin, Maltodextrin, Sodium Saccharin, Helianthus Annuus Seed Oil, Potassium Sorbate, BHT, Limonene, CI 16255.
  Interventions: Drug: Dental foam "Biorepair PERIBIOMA"
- Dental foam "WATER:DENT" (Experimental): Aqua, Xylitol, PVP, PEG-40 Hydrogenated Castor Oil, Hippophae Rhamnoides Extract, Chamomilla Recutita Extract, Sodium Benzoate, Sodium Lauryl Sulfate, Aroma, Propylene Glycol, Olaflur, Potassium Sorbate, Sodium Phosphate, Disodium Phosphate, Menthol, Bisabolol, Menthyl Lactate, PPG-26 Buteth-26, Sodium Saccharin, Sodium Methylparaben, Citric Acid, Limonene.
  Interventions: Drug: Dental foam "WATER:DENT"
- Spray "BUCCOTHERM" (Experimental): Aqua (Castéra-Verduzan Thermal Spring water), Alcohol, Xylitol, Glycerin, Camellia sinensis leaf water, Mentha piperita leaf water, Hydrogenated starch hydrolysate, Aqua, Aroma, Limonene, Benzyl alcohol, Dehydroacetic acid.
  Interventions: Drug: Dental spray "BUCCOTHERM"

INTERVENTIONS:
Other: No intervention (negative control) — The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds.
  Arms: No intervention (negative control)
Other: Water (positive control) — The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds. Then, participants will to rinse their mouth with tap water 60 seconds.
  Arms: Water (positive control)
Drug: Dental foam "Biorepair PERIBIOMA" — The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds.
  Then, participants will use a dental foam "Biorepair PERIBIOMA" to rinse their mouth. They should rinse their mouth for 60 seconds and then spit out the foam.
  Arms: Dental foam "Biorepair PERIBIOMA"
Drug: Dental foam "WATER:DENT" — The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds.
  Then, participants will use a dental foam "WATER:DENT" to rinse their mouth. They should rinse their mouth for 60 seconds and then spit out the foam.
  Arms: Dental foam "WATER:DENT"
Drug: Dental spray "BUCCOTHERM" — The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds.
  Then, participants will use a dental spray "BUCCOTHERM" to rinse their mouth. They should rinse their mouth for 60 seconds and then spit out the foam.
  Arms: Spray "BUCCOTHERM"

SUMMARY:
The aim of the study is to assess the effect of oral foams on salivary pH changes after Coca-cola consumption in young adults.

DETAILED DESCRIPTION:
This will be a cross-over clinical trial assessing the effect of oral foams containing zink hydroxiapatite and probiotics (Lactobacillus, Bifidobacterium), Olaflur (amino fluoride), and oral spray with alkaline thermal water. The study will be conducted in six visits over a period of 1.5 months. After enrolment, dental examination will be performed using the following indices: DMFT, OHI-S index, Bleeding index. Saliva buffer capacity, salivary flow rate, and baseline salivary pH will be measured. Salivary pH changes will be registered after consumption of Coca-cola alone or followed by each of the tested products application.

ELIGIBILITY:
Inclusion Criteria:

* Females and males
* Aged between 18-44 years
* Willingness to comply with all study procedures and availability for the duration of the study.
* Subjects who signed informed consent

Exclusion Criteria:

* History of chemotherapy or radiotherapy;
* An oral mucosa pathology;
* Orthodontic treatment within the previous 3 months;
* Dental bleaching within the previous 3 months;
* Withdrawal of consent;
* Patient refusal to continue participation in the study;
* Detection of an allergic reaction to any components of the dental foams or carbonated drinks used in the study.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
The time required for salivary pH recovery after Coca-Cola consumption | 1 hour
  The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds. They will be asked to spit saliva into a sterile vial at baseline (before Coca-cola consumption), immediately after Coca-Cola consumption and further every 5 minutes until the pH reaches baseline levels. Salivary pH levels will be measured with a digital pH meter. The time required for pH recovery will be registered.
The time required for salivary pH recovery after Coca-Cola consumption followed by oral sprays application | 1 hour
  The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds. Then, participants will be asked to rinse their mouths with tap water (control) or each of the tested oral foams according to the manufacturer's recommendations. They will be asked to spit saliva into a sterile vial at baseline (before Coca-cola consumption), immediately after Coca-Cola consumption, immediately after oral foams/tap water rinse and further every 5 minutes until the pH reaches baseline levels. The pH levels will be measured with a digital pH meter. The time required for pH recovery will be registered.
Minimal value of salivary pH after Coca-Cola consumption | 1 hour
  The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds. They will be asked to spit saliva into a sterile vial at baseline (before Coca-cola consumption), immediately after Coca-Cola consumption and further every 5 minutes until the pH reaches baseline levels. Salivary pH levels will be measured with a digital pH meter. The minimal pH value will be registered.
minimal value of salivary pH recovery after Coca-Cola consumption followed by oral sprays application | 1 hour
  The participants will be asked to hold 20 ml of "coca-cola" in their mouth for 30 seconds. Then, participants will be asked to rinse their mouths with tap water (control) or each of the tested oral foams according to the manufacturer's recommendations. They will be asked to spit saliva into a sterile vial at baseline (before Coca-cola consumption), immediately after Coca-Cola consumption, immediately after oral foams/tap water rinse and further every 5 minutes until the pH reaches baseline levels. The pH levels will be measured with a digital pH meter. The minimal pH value will be registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Dentistry of Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polyakova M, Egiazaryan A, Doroshina V, Zaytsev A, Malashin A, Babina K, Novozhilova N. The Effect of Oral Care Foams and a Spray on Salivary pH Changes after Exposure to Acidic Beverages in Young Adults. Dent J (Basel). 2024 Apr 3;12(4):93. doi: 10.3390/dj12040093. PMID 38668005